CLINICAL TRIAL: NCT05009550
Title: Effect of Erector Spina Plain (ESP) Block on Patient Outcomes in Patients With Liver Tumor Undergoing Radiofrequency Ablation
Brief Title: ESP Block on Patient Outcomes in Patients With Liver Tumor Undergoing Radiofrequency Ablation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Özlem ÖZ GERGİN, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/346
Record Dates: First submitted 2021-08-16; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Hepatic Carcinoma
Keywords: Erector spinae block; Radiofrequency ablation; Hepatocellular Carcinomas; ultrasound
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant
Masking Description: single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block group (ESP) (Active Comparator): Single-shot ultrasound guided ESP block is performed at the T8 vertebral level before the procedure to all patients in ESP block Group. Then standard sedation method is applied to all patients.
  Interventions: Procedure: Group ESP
- Control Group (Other): This Group was received no intervention.Standard sedation method is applied to all patients.
  Interventions: Other: Non-blocked Group

INTERVENTIONS:
Procedure: Group ESP — Single-shot ultrasound guided ESP block is performed at the T8 vertebral level before the procedure to all patients in ESP block Group
  Arms: Erector spinae plane block group (ESP)
Other: Non-blocked Group — This Group is received no intervention.Patients will be sedated as standard and radiofrequency procedure will be applied.
  Arms: Control Group

SUMMARY:
To evaluate the ability of Erector spina Plane Block decrease postoperative pain and analgesia requirements in patients undergoing percutaneous Radiofrequency ablation of Hepatocellular Carcinomas.

DETAILED DESCRIPTION:
Erector spina Plane Block is performed with guided ultrasound at T8 transverse process level lead to adequate intraprocedural and postoperative analgesia, in percutaneous Radiofrequency ablation of Hepatocellular Carcinomas.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients

Exclusion Criteria:

* history of allergy to the study medication
* refused to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Scale assesment | 24 hours after procedure
  A research assistant, blinded to the group allocation, interviewed patients and collected data at 6 times intervals (0.,2.,4.,6.,12 and 24 hours) in the 24 hours postprocedure. Patients will be asked to rate their pain using Numeric Pain Scale, where 0=no pain and 10=worst pain possible.

SECONDARY OUTCOMES:
Demographic data | 24 hours after procedure
  Age, BMI, ASA, Duration of procedure are recorded.
Incidences of adverse effects (like nausea and vomiting) | 24 hours after procedure
  Incidences of adverse effects (like nausea and vomitting) during the 24 hours postprocedure perİod is recorded at 6 times intervals (0,2,4,6,12,24 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Oz Gergin, MD, Principal Investigator — TC Erciyes University
Locations (1):
- Özlem Öz Gergin, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De- identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be available within 24 months of study completion
Access Criteria: Data accept requests will be reviewed by an external independent Review Panel.Requesters will be required to sign a Data Access Agreement.

REFERENCES:
- [Result] Wells SA, Hinshaw JL, Lubner MG, Ziemlewicz TJ, Brace CL, Lee FT Jr. Liver Ablation: Best Practice. Radiol Clin North Am. 2015 Sep;53(5):933-71. doi: 10.1016/j.rcl.2015.05.012. PMID 26321447
- [Result] Joung KW, Choi SS, Jang DM, Kong YG, Lee HM, Shim JH, Won HJ, Shin YM, Kim PN, Song MH. Comparative Effects of Dexmedetomidine and Propofol on US-Guided Radiofrequency Ablation of Hepatic Neoplasm Under Monitored Anesthesia Care: A Randomized Controlled Study. Medicine (Baltimore). 2015 Aug;94(32):e1349. doi: 10.1097/MD.0000000000001349. PMID 26266387